CLINICAL TRIAL: NCT05024110
Title: Response of Vitamin D and Parathormone to Different Exercise Intensities in Children With Down's Syndrome: a Clinical Controlled Trial
Brief Title: Effect of Exercise Intensity on Vitamin D
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taif University (Other)
Responsible Party: Principal Investigator, Hatem Allam, Assistant Prof., Taif University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 428
Record Dates: First submitted 2021-08-23; First posted 2021-08-27 (Actual); Last update posted 2021-09-01 (Actual); Status verified 2021-08

CONDITIONS: Down Syndrome; Vitamin D Deficiency
MeSH Terms: conditions — Down Syndrome; Vitamin D Deficiency

STUDY DESIGN:
Intervention Model Description: A randomized controlled trial was used to investigate the effect of exercise intensity on vitamin D and PTH levels in children with Down's syndrome. The enrollment of the participants was done by telephone calls to their parents or legal guardians. A total of fifty male DS subjects were initially selected to participate in the study. Only forty-four subjects completed the interventional study because six children were excluded. three children did not meet the inclusion criteria, parents of two children refused to complete the study, and one lost to follow-up. Their age was ranged from 8-12 years. The participants were assigned randomly using sealed envelopes into two equal groups; group I (GI) and group II (GII) each contain twenty-two subjects. GI received the high-intensity T-AE and the GII received the moderate-intensity T-AE, three times per week for three months. All subjects were selected from hospitals in the Western area, Saudi Arabia.
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (Experimental): GI received high-intensity exercise training.
  Interventions: Other: High intensity treamill exercise training.
- Group II (Experimental): GII received moderate-intensity exercise training.
  Interventions: Other: Moderate intensity treamill exercise training.

INTERVENTIONS:
Other: High intensity treamill exercise training. — We used the Martti Karvonen formula to calculate the heart rate zone. Firstly, the resting heart rate (rest-HR) was detected for every participant by inviting him to lie in a prone position for 10 minutes while catching a heart rate monitor. After that, the maximum heart rate (max-HR) was calculated by utilizing this formula: maximum heart rate =220- age. Then, we calculated the heart rate reserve (HRR) by using the law: HRR= max-HR - resting HR. Exercise intensity is represented as a percentage of HRR. Finally, the target heart rate (target-HR) was calculated by using the formula: target-HR = HRR x intensity% + rest-HR. Moderate-intensity exercises are defined as the activity which uses 50% to 70% of the HRR, while high-intensity exercises use 70% to 90% of the HRR
  Arms: Group I
Other: Moderate intensity treamill exercise training. — We used the Martti Karvonen formula to calculate the heart rate zone. Firstly, the resting heart rate (rest-HR) was detected for every participant by inviting him to lie in a prone position for 10 minutes while catching a heart rate monitor. After that, the maximum heart rate (max-HR) was calculated by utilizing this formula: maximum heart rate =220- age. Then, we calculated the heart rate reserve (HRR) by using the law: HRR= max-HR - resting HR. Exercise intensity is represented as a percentage of HRR. Finally, the target heart rate (target-HR) was calculated by using the formula: target-HR = HRR x intensity% + rest-HR. Moderate-intensity exercises are defined as the activity which uses 50% to 70% of the HRR, while high-intensity exercises use 70% to 90% of the HRR
  Arms: Group II

SUMMARY:
Children with Down's syndrome (DS) are more liable to vitamin D deficiency. Treating this deficiency with supplements is associated with the risk of intoxication due to increased intestinal absorption or decreased vitamin D metabolism. The aim of the study was to compare the effect of two exercise intensities on the modulation of vitamin D and Parathormone (PTH) levels in children with DS.

DETAILED DESCRIPTION:
Forty-four DS male children aged from 8-12 years participated in the study. The subjects were assigned randomly into two equal groups. group I received high-intensity treadmill aerobic exercises (T-AE) and group II received moderate-intensity T-AE, three times per week for three months. the blood samples were collected from both groups before the intervention, after one month of intervention, then after three months of intervention to assess serum 25(OH)D and PTH levels.

ELIGIBILITY:
Inclusion Criteria:

* all subjects were trainable and able to walk freely without assistance.
* Had vitamin D deficiency, the serum level of 25-hydroxyvitamin D (25(OH) D) was ranged from 10-20ng/mL.
* Did not take calcium or vitamin D3 supplements, medications for osteoporosis, antiepileptic drugs, or any medications that may affect the vitamin D metabolism in the last 5 months.
* The feeding method during the first two years of age for all children was bottle feeding.
* Mild to moderate mentally retarded, (IQ ranged from 45-70) to be able to understand and obey simple orders.
* free from any medical consequences for example cardiopulmonary disorders, auditory defects, and visual impairments.
* Had no previous history of strength training.
* Body mass index percentile ranged from the 50th percentile to less than the 75th percentile (healthy).
* The feeding method was by mouth with no special diet, with an absence of signs of malnutrition

Exclusion Criteria:

* autoimmune disease.
* Renal diseases.
* Have taken any thyroid medications.
* Obesity.
* epileptic fits.

Ages: 8 Years to 12 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes — All children were male
Enrollment: 44 (Actual)
Dates: Start 2021-01-25 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-05-14 (Actual)

PRIMARY OUTCOMES:
vitamin d after one month | one month
  serum level of 25(OH) D ng/ml after one month of intervention
vitamin d after three months | three months
  serum level of 25(OH) D ng/ml after three months of intervention
PTH after one month | one month
  Serum level of parathormone (PTH) pmol/L after one month of intervention
PTH after three months | three months
  Serum level of parathormone (PTH) pmol/L after three months of intervention

CONTACTS AND LOCATIONS:
Locations (1):
- College of applied medical sciences, Ta'if, Mecca Region, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No